CLINICAL TRIAL: NCT03263442
Title: Randomized Placebo Controlled Trial of High Dose Intravenous Thiamine for the Prevention of Delirium in Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: High Dose Intravenous Thiamine for the Prevention of Delirium in Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LCCC1726; CCR-17-300 (Other Grant/Funding Number: Rising Tide Foundation for Clinical Cancer Research)
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Hematopoietic Stem Cell Transplantation; Delirium; Thiamine Deficiency
MeSH Terms: conditions — Delirium; Thiamine Deficiency | interventions — Thiamine; thiamine hydrochloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Thiamine 200 mg IV
  Interventions: Drug: Thiamine
- Control (Placebo Comparator): Normal saline IV
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Thiamine — 200 mg IV three times daily for seven days
  Other Names: Thiamine Hydrochloride Injection
  Arms: Intervention
Drug: Normal saline — Normal saline IV three times daily for seven days
  Other Names: Placebo
  Arms: Control

SUMMARY:
Purpose: To conduct a randomized controlled pilot study investigating the use of high dose intravenous (IV) thiamine to prevent delirium and mitigate the long-term effects of delirium, including health-related quality of life (HRQOL), functional status, and neuropsychiatric outcomes, in patients admitted to University of North Carolina (UNC) Hospital for allogeneic hematopoietic stem cell transplant (HSCT).

Participants: 60 adult inpatients admitted to the UNC Bone Marrow Transplant Unit for allogeneic stem cell transplant.

Procedures (methods): Participants will be admitted for allogeneic HSCT and on the day after transplant randomized to seven days of high dose IV thiamine or placebo. Thiamine levels will be measured weekly and participants will be assessed for evidence of delirium using validated measures. Validated measures will also be used to assess cognitive function, depression, post-traumatic stress symptoms, functional status, and HRQOL prior to hospitalization and at one, three, and six months after transplant.

DETAILED DESCRIPTION:
Delirium is a common and potentially preventable neuropsychiatric complication in cancer patients receiving hematopoietic stem cell transplantation (HSCT) that has profound consequences. Among cancer patients hospitalized for HSCT, delirium occurs in approximately 40% of patients and increases the risk of mortality. Long-term, delirium in this population results in worse physical health, mental health, and quality of life. Though strategies to prevent delirium have the potential to significantly improve the lives of people living with cancer, research in this area is extremely limited. Thiamine deficiency is also ubiquitous during HSCT and a known contributor to the development of delirium in other patient populations. High dose intravenous (IV) thiamine is an evidence-based and promising treatment for delirium, but no one has studied IV thiamine as a prevention strategy.

This is a randomized double-blind controlled trial in participants undergoing allogeneic HSCT to determine if high dose IV thiamine can prevent delirium and minimize the deleterious impact of delirium on health-related quality of life (HRQOL), functional status, and other neuropsychiatric outcomes. The investigators will recruit 60 patients admitted for allogeneic HSCT at UNC, randomize them to treatment with high dose IV thiamine (n = 30) versus placebo (n = 30), and systematically evaluate all participants for delirium and related comorbidities. The investigators will use the Delirium Rating Scale (DRS) to measure the severity and duration of delirium immediately prior to transplant and after HSCT until 30 days post-transplant or discharge. If delirium is identified, the DRS will be administered daily until delirium resolves. The investigators will obtain thiamine levels and other laboratory parameters associated with delirium the day after transplant, and continue to monitor thiamine levels weekly thereafter. The investigators will also monitor HRQOL, functional status, depression, post-traumatic stress symptoms, and cognitive function prior to transplant and at one, three, and six months after transplant to elucidate the persistent impact of delirium in this population and the potential for thiamine to mitigate these negative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the UNC Hospital Bone Marrow Transplant Unit for allogeneic stem cell transplant
* At least 18 years of age
* Able to speak English
* Able to provide informed consent

Exclusion Criteria:

* A history of adverse reaction to IV thiamine
* Pregnancy, confirmed by a negative pregnancy test within 30 days of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Rosenstein, MD, Study Chair — University of North Carolina, Chapel Hill; Zev Nakamura, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nakamura ZM, Deal AM, Park EM, Quillen LJ, Chien SA, Stanton KE, McCabe SD, Heiling HM, Wood WA, Shea TC, Rosenstein DL. A randomized double-blind placebo-controlled trial of intravenous thiamine for prevention of delirium following allogeneic hematopoietic stem cell transplantation. J Psychosom Res. 2021 Jul;146:110503. doi: 10.1016/j.jpsychores.2021.110503. Epub 2021 Apr 27. PMID 33945982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the UNC Bone Marrow Transplant and Cellular Therapies Unit from October 2017 through February 2020.
Pre-assignment Details: Of the 66 participants who enrolled in the study, 2 withdrew prior to randomization.
Period: Inpatient Phase
Arm/Group | Intervention | Control
Started | 30 | 34
Completed | 28 | 33
Not Completed | 2 | 1
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Inadequate Drug Exposure | 0 | 1
Period: 1-month Follow-Up
Arm/Group | Intervention | Control
Started | 28 | 33
Completed | 27 | 33
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: 3-month Follow-Up
Arm/Group | Intervention | Control
Started | 27 | 33
Completed | 26 | 30
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3
Period: 6-month Follow-Up
Arm/Group | Intervention | Control
Started | 26 | 30
Completed | 24 | 28
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: Only participants who met the following a priori criteria were counted: 1.) received all seven days of the treatment; 2.) received at least 17/21 (80%) scheduled study drug doses; and 3.) delirium was assessed at least weekly until the participant was found to be delirious, reached 30 days post-transplant, or was discharged.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 28 | 33 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (12.5) | 53.6 (14.7) | 54.2 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 17 | 20 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 27 | 32 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 25 | 27 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 33 | 61
Education [Mean (Standard Deviation); unit: years] — Years of education
  years | 14.7 (2.7) | 15.3 (2.7) | 15.0 (2.7)
Diagnosis [Count of Participants; unit: Participants]
  Acute leukemia | 18 | 19 | 37
  Chronic leukemia | 2 | 5 | 7
  Lymphoma | 0 | 2 | 2
  Myelodysplastic Syndrome | 5 | 5 | 10
  Myeloproliferative Disorder | 2 | 1 | 3
  Other | 1 | 1 | 2
CIBMTR Disease Risk Index [Count of Participants; unit: Participants] — CIBMTR: Center for International Blood and Marrow Transplant Research. Uses disease, stage, and cytogenetics to assigns low, intermediate, high, or very high risk related to overall survival after allogeneic hematopoietic stem cell transplant among patients with hematologic malignancies.
  Participants
    N/A | 3 | 3 | 6
    low | 17 | 19 | 36
    intermediate | 3 | 9 | 12
    high | 5 | 2 | 7
Donor Type [Count of Participants; unit: Participants]
  Matched Related Donor | 9 | 10 | 19
  Matched Unrelated Donor | 16 | 18 | 34
  Haploidentical | 3 | 5 | 8
Conditioning Regimen [Count of Participants; unit: Participants]
  Myeloablative | 15 | 13 | 28
  Reduced Intensity or Non-Myeloablative | 13 | 20 | 33
ECOG Score [Count of Participants; unit: Participants] — A scale by the Eastern Cooperative Oncology Group (ECOG) from 0-5 to describe patient's selfcare ability and activity level.
  0, Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 13 | 18 | 31
    1 | 15 | 14 | 29
    2 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Delirium
Description: Delirium incidence will be measured using the Delirium Rating Scale (DRS). The DRS is a is a 10-item, clinician-rated scale that rates the severity of delirium symptoms over a 24-hour period using all available information from the patient interview, mental status examination, medical history and tests, nursing observations, and family reports. The maximum possible score is 32. Higher scores suggest more severe symptoms. A cut-off score of > 12 has been suggested to distinguish patients with delirium from patients with other neuropsychiatric disorders. Delirium incidence will be defined as at least one assessment with DRS > 12.
Time Frame: Assessments will occur in the week prior to transplant, then 3 times weekly post-transplant until 30 days post-transplant or discharge, whichever comes first.
Population: The analysis population was defined a priori as those participants who: 1.) received at least 17 of 21 (80%) scheduled study drug doses; 2.) received at least one dose on each of the study drug administration days; and 3.) had no fewer than one DRS assessment per week until they were found to be delirious, reached 30 days post-transplant, or were discharged.
Measure: Number; unit: percentage of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 33
percentage of participants | 25 | 21

2. Secondary Outcome: Delirium Severity
Description: Delirium severity will be measured using the Delirium Rating Scale (DRS). The DRS is a is a 10-item, clinician-rated scale that rates the severity of delirium symptoms over a 24-hour period using all available information from the patient interview, mental status examination, medical history and tests, nursing observations, and family reports. The score ranges from 0 to 32 with higher scores reflecting more severe symptoms. A cut-off score of > 12 has been suggested to distinguish patients with delirium from patients with other neuropsychiatric disorders. The DRS medians and ranges are reported for each group at baseline and in each week of hospitalization for thiamine and placebo groups.
Time Frame: Assessments will occur in the week prior to transplant (baseline), then at least 3 times post-transplant on a weekly basis until 30 days post-transplant or discharge, whichever comes first, up to week 5
Population: Attrition over time is due to hospital discharge (primary reason), withdrawal, or death.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 33
score on a scale
  Baseline | 4.0 [2.0 to 8.0] | 4.0 [2.0 to 7.0]
  Week 1 | 4.83 [3.0 to 9.0] | 4.67 [2.67 to 15.00]
  Week 2: number analyzed (Participants) | 28 | 32
  Week 2 | 6.50 [2.67 to 20.33] | 5.33 [2.33 to 16.00]
  Week 3: number analyzed (Participants) | 23 | 26
  Week 3 | 6.33 [1.00 to 18.60] | 5.17 [2.00 to 17.80]
  Week 4: number analyzed (Participants) | 7 | 7
  Week 4 | 5.50 [4.00 to 20.00] | 6.00 [5.00 to 13.50]
  Week 5: number analyzed (Participants) | 1 | 4
  Week 5 | 20.00 [20.00 to 20.00] | 7.50 [4.00 to 8.00]

3. Secondary Outcome: Delirium Duration
Description: Delirium duration will be measured using the Delirium Rating Scale (DRS). The DRS is a is a 10-item, clinician-rated scale that rates the severity of delirium symptoms over a 24-hour period using all available information from the patient interview, mental status examination, medical history and tests, nursing observations, and family reports. The maximum possible score is 32. Higher scores suggest more severe symptoms. A cut-off score of > 12 has been suggested to distinguish patients with delirium from patients with other neuropsychiatric disorders. Delirium duration will be reported as number of consecutive days during which DRS > 12.
Time Frame: as for outcome 1
Population: These analyses are exclusive to those participants who experienced delirium.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 7 | 7
days | 2.0 (1.2) | 4.4 (4.7)

4. Secondary Outcome: Concentration of Thiamine Status Stratified by Delirium Status
Description: The relationship between thiamine levels at the end of the seven day administration of thiamine and the development of delirium at any point during the thirty days post-transplant or the post-transplant hospitalization, whichever comes first, will be examined. Thiamine levels (nmol/L) are presented in participants who did and did not experience delirium.
Time Frame: From end of 7-day intervention period until the development of delirium at any point during the post-transplant hospitalization up to a maximum of 30 days
Population: Only those participants in whom thiamine levels were obtained at the end of the seven day administration were included.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Delirium: Participants who experienced delirium, defined as at least one DRS score >12, during the post-transplant hospitalization.
- No Delirium: Participants who did not meet criteria for delirium during the post-transplant hospitalization.
Arm/Group | Delirium | No Delirium
Number analyzed (Participants) | 14 | 45
nmol/L | 115.6 (69.3) | 93.8 (28.5)

5. Secondary Outcome: Change in Health-related Quality of Life Scores (Month 1)
Description: HRQOL will be assessed using the Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT). The FACT-BMT is a 47-item self-administered assessment which asks individuals to rate questions related to physical, social/family, emotional, and functional well-being on a 5-point Likert Scale (0, not at all to 4, very much). Scores are summed across the items, resulting in a score from 0 to 148, with higher scores indicating better quality of life. Negative change scores indicate worse HRQOL with time.
Time Frame: From baseline to one month post-transplant
Population: Participants who completed the 1 month follow-up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 33
score on a scale | -7.53 (11.66) | -5.69 (11.59)

6. Secondary Outcome: Change in Health-related Quality of Life Scores (Month 3)
Description: as for outcome 5
Time Frame: Baseline to three months post-transplant
Population: Participants who completed the 3 month follow-up period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 30
score on a scale | -3.96 (9.11) | -1.43 (16.79)

7. Secondary Outcome: Change in Health-related Quality of Life Scores (Month 6)
Description: as for outcome 5
Time Frame: Baseline to six months post-transplant
Population: Participants who completed the 6 month follow-up period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
score on a scale | -4.36 (14.09) | 0.28 (12.17)

8. Secondary Outcome: Change in Depression Scores (Month 1)
Description: Depression will be assessed using the Patient Reported Outcomes Measurement Information System - Depression (PROMIS-D) 8a short form. Scores for all PROMIS measures are reported on the T-score metric in which the mean=50 and standard deviation (SD) = 10 are centered on the general population means. Higher scores represent greater degrees of mood symptoms. Positive change scores indicate worse mood over time.
Time Frame: Baseline to one month post-transplant
Population: Participants who completed the 1 month follow-up period.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 33
T-score | -1.34 (8.28) | 1.16 (6.12)

9. Secondary Outcome: Change in Depression Scores (Month 3)
Description: as for outcome 8
Time Frame: Baseline to three months post-transplant
Population: Participants who completed the 3 month follow-up period
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 30
T-score | 0.93 (6.24) | 0.32 (9.53)

10. Secondary Outcome: Change in Depression Scores (Month 6)
Description: as for outcome 8
Time Frame: Baseline to six months post-transplant
Population: Participants who completed the 6 month follow-up period
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
T-score | 0.14 (6.88) | -1.66 (7.89)

11. Secondary Outcome: Change in Post-traumatic Stress Symptom Scores (Month 1)
Description: Post-traumatic stress symptoms will be measured using the Post Traumatic Stress Syndrome Scale 14 (PTSS-14). The PTSS-14 is a 14-item self-administered assessment. Questions are on a 7-point Likert-type Scale (1, never to 7, always) resulting in a total score between 14 and 98. Higher scores represent a more likely diagnosis of post-traumatic stress disorder (PTSD). Positive change scores indicate worse post-traumatic stress over time.
Time Frame: Baseline to one month post-transplant
Population: Participants who completed the 1 month follow-up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 33
score on a scale | -0.52 (10.88) | 1.55 (6.92)

12. Secondary Outcome: Change in Post-traumatic Stress Symptom Scores (Month 3)
Description: as for outcome 11
Time Frame: Baseline to three months post-transplant
Population: Participants who completed the 3 month follow-up period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 30
score on a scale | -1.50 (6.58) | 0.83 (5.63)

13. Secondary Outcome: Change in Post-traumatic Stress Symptom Scores (Month 6)
Description: as for outcome 11
Time Frame: Baseline to six months post-transplant
Population: Participants who completed the 6 month follow-up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
score on a scale | 1.79 (9.14) | 1.32 (7.00)

14. Secondary Outcome: Change in Cognitive Function Scores (Month 1)
Description: Cognitive function will be assessed using the Montreal Cognitive Assessment (MOCA). The MOCA is a clinician-administered tool with scores ranging from 0 to 30. Lower scores indicate worse cognitive function. Scores ≤ 25 are considered clinically significant. Positive change scores indicate better function with time.
Time Frame: From baseline to one month post-transplant
Population: One participant in the control arm was unable to complete the MoCA due to restrictions on in-person human subjects research during the COVID-19 pandemic. Otherwise, all participants available at the 1-month follow-up time point were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 32
score on a scale | -0.70 (3.35) | -0.09 (2.76)

15. Secondary Outcome: Change in Cognitive Function Scores (Month 3)
Description: as for outcome 14
Time Frame: Baseline to three months post-transplant
Population: Participants who completed the 3 month follow-up period and we able to participate in the cognitive assessment. Of the 26 participants active in the thiamine arm at the 3 month follow-up, 1 did not complete this measure due to barriers related to the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 30
score on a scale | -0.12 (0.97) | 0.97 (2.82)

16. Secondary Outcome: Change in Cognitive Function Scores (Month 6)
Description: as for outcome 14
Time Frame: From baseline to six months post-transplant
Population: Participants who completed the 6 month follow-up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
score on a scale | 0.71 (3.32) | 1.54 (2.87)

17. Secondary Outcome: Change in Functional Status Scores (Month 1)
Description: Functional status will be measured using the Eastern Cooperative Oncology Group (ECOG) performance scale. ECOG performance status is a single question scored on a 6-point scale (range 0 to 5) with higher scores representing greater physical restriction due to illness. Negative change scores indicate better function with time.
Time Frame: Baseline to one month post-transplant
Population: Participants who completed the 1 month follow-up period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 27 | 33
score on a scale | 0.70 (0.67) | 0.88 (0.93)

18. Secondary Outcome: Change in Functional Status Scores (Month 3)
Description: as for outcome 17
Time Frame: From baseline to three months post-transplant
Population: Participants who completed the 3 month follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 26 | 30
score on a scale | 0.69 (0.62) | 0.60 (0.89)

19. Secondary Outcome: Change in Functional Status Scores (Month 6)
Description: as for outcome 17
Time Frame: Baseline to six months post-transplant
Population: Participants who completed the 6 month follow-up period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 24 | 28
score on a scale | 0.46 (0.93) | 0.21 (0.63)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were only collected from October 2017 through February 2020, during the intervention phase of the study and coinciding with participants' hospitalization for hematopoietic stem cell transplantation. This phase lasted up to 30 days for each participant. The study was completed on August 10, 2020, as secondary outcomes were collected for an additional 5 months after completion of AE data collection.
Description: Adverse events were were graded per NCI CTCAE v. 4 criteria.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/34
Other Adverse Events (participants affected / at risk) | 0/30 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03263442/Prot_SAP_000.pdf